CLINICAL TRIAL: NCT04956913
Title: Macintosh Versus Macgrath for Laryngoscopy in COVID 19 Hypoxemic ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of anesthesia and intensive care department, Mongi Slim Hospital
Other Study IDs: macintosh versus Mac Grath
Record Dates: First submitted 2021-07-08; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: Tracheal intubation; mechanical ventilation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mac Grath: Patients of this group were intubated using Mac Gath videolaryngoscope
  Interventions: Device: Mac Grath
- Machintosh: Patients of this group were intubated using the classic Macintosh laryngscoscope
  Interventions: Device: Macintosh

INTERVENTIONS:
Device: Mac Grath — Patients of this group were intubated using Mac Gath videolaryngoscope
  Groups: Mac Grath
Device: Macintosh — Patients of this group were intubated using the Macintosh Laryngoscope
  Groups: Machintosh

SUMMARY:
In this comparative prospective study, we aim to compare the classic Macintosh laryngoscope and the Mac Grath videolaryncoscope in ICU covid 19 patients recruiting intubation and invasive mechanical ventilation.

patients meeting inclusion criteria were randomized in 2 groups: MacGrath and Macintosh.

we collected anthropometric and intubation data among all patients, and the 2 groups were compared regarding the time for intubation, the need of alternative techniques to intubate and the impact on the oxygenation by recording the lowest SPO2.

DETAILED DESCRIPTION:
In this comparative prospective study, we aim to compare the classic Macintosh laryngoscope and the Mac Grath videolaryncoscope in ICU covid 19 patients recruiting intubation and invasive mechanical ventilation.

All hypoxemic COVID19 patients requiring intubation were enrolled in this trial.

all patients had a preoxygenation with non invasive ventilation with 100% oxygen.

patients meeting inclusion criteria were randomized in 2 groups: MacGrath and Macintosh.

we collected anthropometric and intubation data among all patients, and the 2 groups were compared regarding the time for intubation, the need of alternative techniques to intubate and the impact on the oxygenation by recording the lowest SPO2.

ELIGIBILITY:
Inclusion Criteria:

* All COVID 19 hypoxemic patients requiring tracheal intubation

Exclusion Criteria:

* hypoxemic cardiac arrest before intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU covid 19 patients requiring tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Time for tracheal intubation | 10 minutes
  Time from the blade pass the lips until the first breath was administred

IPD SHARING:
Plan to Share IPD: No